CLINICAL TRIAL: NCT00358514
Title: Continuous Compartment Pressure Monitoring (Ccpm) Following Tibial Fracture: A Prospective Randomized Trial
Brief Title: Continuous Pressure Monitoring In Lower Leg Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Large sample size and change in Orthopaedic practice to use of CCPM in conjunction with Clinical Monitoring rendered project less timely.
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. P.J. O'Brien, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C06-0063
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Compartment Syndrome
Keywords: Tibia; fracture; compartment syndrome; fasciotomy
MeSH Terms: conditions — Compartment Syndromes; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Continuous Compartment Pressure Monitoring — See Detailed Description.

SUMMARY:
This study has been designed to allow us to learn more about diagnosing Compartment Syndrome, which is a condition that occurs in approximately 5% of tibial (lower leg) fractures. In Compartment Syndrome, nerves, muscle and blood vessels are affected by swelling within the enclosed spaces (compartments) of the leg. The tissue covering these compartments (called the fascia) is not expandable and is not able to accommodate this swelling, and so the tissues within the compartments become compressed. If the pressure is not relieved it can result in blood flow being blocked to the inside of the compartment (muscle, blood vessels, and nerves) which can lead to permanent injury to the muscle and nerves. Late complications in untreated compartment syndrome include a failure of the injured bone to heal, nerve damage, and contracture (shortening) of muscle, all of which can result in a weak, painful, stiff, and poorly formed limb that is not functioning well, and could result in amputation.

DETAILED DESCRIPTION:
This study has been designed to prospectively evaluate the clinical results of the use of Continuous Compartment Pressure Monitoring (CCPM) in the treatment of tibial fractures.

Fractures of the tibia cause local haemorrhage, tissue edema and swelling within the indistensible fascial compartments of the leg. In a proportion of patients, pressure within the compartments rises sufficiently high to reduce capillary bed perfusion, resulting in tissue ischemia. This condition is termed compartment syndrome and complicates approximately 5% tibial fractures. The early and late morbidity from untreated compartment syndrome is important. In the early period, severe pain, local muscle necrosis and infection may occur, and systemically, rhabdomyolysis may result in renal failure. Multiple surgical procedures and a prolonged period of hospital treatment may be required to address these complications. Ultimately the affected limb may loose viability and require amputation. Later, non-union of bone, contracture of muscle and permanent nerve palsy may result in a limb that is painful, deformed, weak and stiff with dystrophic and vulnerable skin. This may result in functional impairment, loss of employment, or again amputation.

The treatment of compartment syndrome by emergency fasciotomy of all four leg compartments is universally accepted. However, there is a small but significant level of morbidity associated with this procedure. Local cutaneous nerves may be inadvertently divided, the open wounds may become infected, and the staged closure of such wounds may require several operative procedures under general anaesthetic. The resulting scars are cosmetically prominent and unsightly, and may be hypersensitive or fragile.

The diagnosis of compartment syndrome may be problematic. The clinical features are well described, but in the individual patient may be equivocal, atypical, or masked by analgesia or obtunded consciousness. Although cases of acute compartment syndrome are very rarely missed altogether in contemporary practice, the diagnosis can be delayed for many hours because of uncertainty or lack of awareness of the importance of a subtle and evolving clinical picture. This delay in diagnosis exposes the patient to prolonged compartmental ischemia and an increased risk of complications.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age and older, presenting for treatment in 24 hours or less
* Diaphyseal or bicondylar plateau fracture of the tibia

Exclusion Criteria:

* Patients under 16 years of age
* Patients who present to VGH more than 24 hours after the injury
* Patients who are not mentally competent to give Informed Consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Outcome measures will be assessed at the time of discharge and at the six and twelve month clinical appointments and will be as follows:
Fasciotomy rate

SECONDARY OUTCOMES:
Outcome measures will be assessed at the time of discharge and at the six and twelve month clinical appointments and will be as follows:Time from injury to fasciotomy 2) Early local outcomes 3) Late local outcomes

CONTACTS AND LOCATIONS:
Overall Officials: P J O'Brien, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada